CLINICAL TRIAL: NCT04737187
Title: An Open-label, Randomized, Phase III Study Comparing Trifluridine/Tipiracil in Combination With Bevacizumab to Trifluridine/Tipiracil Monotherapy in Patients With Refractory Metastatic Colorectal Cancer (SUNLIGHT Study)
Brief Title: Phase III Study of Trifluridine/Tipiracil With and Without Bevacizumab in Refractory Metastatic Colorectal Cancer Patients
Acronym: SUNLIGHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Collaborators: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL3-95005-007; 2020-001976-14 (EudraCT Number)
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Refractory Metastatic Colorectal Cancer
Keywords: trifluridine/tipiracil/lonsurf; TAS102; bevacizumab; avastin; RAS status (wild type, mutant)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trifluridine/Tipiracil + Bevacizumab (Experimental): Participants were administered 35 milligrams per square meter per dose (mg/m²/dose) trifluridine/tipiracil (FTD/TPI) orally twice a day (BID), within 1 hour after completion of morning and evening meals, 5 days on (Day 1 to 5 and Day 8 to 12) with 2 days off (Day 6 to 7 an Day 13 to 14), over 2 weeks, followed by a 14-day rest; with bevacizumab (5 milligrams per kilogram [mg/kg], intravenous [IV] infusion administered every 2 weeks (Day 1 and Day 15). This treatment cycle was repeated every 4 weeks.
  Interventions: Drug: Trifluridine/Tipiracil; Drug: Bevacizumab
- Trifluridine/Tipiracil (Active Comparator): Participants were administered 35 mg/m²/dose of FTD/TPI orally BID, within 1 hour after completion of morning and evening meals, 5 days on (Day 1 to 5 and Day 8 to 12) with 2 days off (Day 6 to 7 and Day 13 to 14), over 2 weeks, followed by a 14-day rest. This treatment cycle was repeated every 4 weeks.
  Interventions: Drug: Trifluridine/Tipiracil

INTERVENTIONS:
Drug: Trifluridine/Tipiracil — Taken by mouth two times a day, 5 days on/2 days off, over 2 weeks, followed by a 14-day rest
  Other Names: TAS102; S 95005; Lonsurf
Drug: Bevacizumab — administered every 2 weeks (Day 1 and Day 15)
  Other Names: Avastin
  Arms: Trifluridine/Tipiracil + Bevacizumab

SUMMARY:
This study is designed as an international, open-label, controlled two-arm, randomized phase III comparison study evaluating the efficacy and safety of trifluridine/tipiracil in combination with bevacizumab versus trifluridine/tipiracil monotherapy in patients with refractory mCRC.

DETAILED DESCRIPTION:
This is an international, open-label, controlled two-arm, randomised phase III study evaluating the efficacy and safety of trifluridine/tipiracil in combination with bevacizumab versus trifluridine/tipiracil monotherapy in patients with refractory mCRC. The analysis will be done after 331 events are reported. In order to observe this number of events, 490 patients will be randomised (1:1) to receive trifluridine/tipiracil in combination with bevacizumab (experimental arm) or trifluridine/tipiracil monotherapy (control arm).

ELIGIBILITY:
Inclusion Criteria:

1. Has histologically confirmed unresectable adenocarcinoma of the colon or rectum (all other histological types are excluded).
2. RAS status must have been previously determined (mutant or wild-type) based on local assessment of tumor biopsy.
3. Has received a maximum of 2 prior chemotherapy regimens for the treatment of advanced colorectal cancer and had demonstrated progressive disease or intolerance to their last regimen.
4. Has measurable or non-measurable disease as defined by RECIST version 1.1
5. Is able to swallow oral tablets.
6. Estimated life expectancy ≥12 weeks.
7. Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1

Exclusion Criteria:

1. More than 2 prior chemotherapy regimens for the treatment of advanced colorectal cancer.
2. Pregnancy, lactating female or possibility of becoming pregnant during the study.
3. Patients currently receiving or having received anticancer therapies within 4 weeks prior to randomization.
4. Has not recovered from clinically relevant non-hematologic CTCAE grade ≥ 3 toxicity of previous anticancer therapy prior to randomization (excluding alopecia, and skin pigmentation).
5. Has symptomatic central nervous system metastases that are neurologically unstable or requiring increasing doses of steroids to control CNS disease.
6. Has severe or uncontrolled active acute or chronic infection.
7. Has active or history of interstitial lung disease and/or pneumonitis, or pulmonary hypertension.
8. Known Hepatitis B or Hepatitis C Virus infection.
9. Known carriers of HIV antibodies.
10. Confirmed uncontrolled arterial hypertension (defined as systolic blood pressure ≥ 150 mm Hg and/or diastolic blood pressure ≥ 100 mm Hg) or uncontrolled or symptomatic arrhythmia.
11. Deep arterial thromboembolic events including cerebrovascular accident or myocardial infarction within the last 6 months prior to randomization.
12. Treatment with any of the following within the specified time frame prior to randomization:

    * major surgery within 4 weeks prior to randomisation (the surgical incision should be fully healed prior to study drug administration), or has not recovered from side effects of previous surgery, or patient that may require major surgery during the study
    * Prior radiotherapy if completed less than 4 weeks before randomisation, except if provided as a short course for symptoms palliation only.
    * Drainage for ascites, pleural effusion or pericardial fluid within 4 weeks prior to randomization
13. Other clinically significant medical conditions.
14. Other malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Tabernero, Prof, Principal Investigator — Vall d'Hebron Institute of Oncology
Locations (99):
- United States (12):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - City of Hope - South Pasedena, South Pasadena, California
  - City of Hope - Upland, Upland, California
  - Mayo Clinic - FL, Jacksonville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Comprehensive Hematology Oncology, St. Petersburg, Florida
  - DuPage Medical Group - Joliet Oncology-Hematology Associates, Joliet, Illinois
  - Investigative Clinical Research of Indiana LLC, Noblesville, Indiana
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Mayo Clinic - Rochester, Rochester, New York
  - Renovatio Clinical - El Paso, El Paso, Texas
- Austria (7):
  - "Medizinische Universität Graz ", Graz
  - "Medizinische Universität Innsbruck Univ.-Klinik für Innere Medizin V", Innsbruck
  - "Ordensklinikum Linz Barmherzige Schwestern Interne I", Linz
  - "Landeskrankenhaus Feldkirch Interne E", Rankweil
  - "Landeskrankenhaus (SALK) Universitätsklinik für Innere Medizin III (SALK)", Salzburg
  - "Allgemeines Krankenhaus - Universitätskliniken Klinische Abteilung für Onkologie", Vienna
  - "Landesklinikum Wiener Neustadt ", Wiener Neustadt
- Belgium (5):
  - "OLV Ziekenhuis Oncology", Aalst
  - "Universitair Ziekenhuis Antwerpen Oncologie", Edegem
  - "UZ Leuven Campus Gasthuisberg Digestieve Oncologie", Leuven
  - "CHC Montlégia Oncologie", Liège
  - "AZ NIKOLAAS Oncology", Sint-Niklaas
- Brazil (6):
  - "Hospital do Câncer de Barretos - Fundação Pio XII Unidade de Pesquisa Clínica", Barretos
  - "Hospital de Base Centro Integrado de Pesquisa", São José do Rio Preto
  - "ICESP - Instituto do Câncer do Estado de São Paulo Centro Integrado de Pesquisa", São Paulo
  - Hospital A C Camargo Unidade de Pesquisa Clinica Rua Antonio Prudente, São Paulo
  - Hospital Sao Camilo Nucleo de Pesquisa Av Alcantara Machado, São Paulo
  - Hospital Albert Einstein Instituto de Ensino e Pesquisa Av Albert Einstein, São Paulo
- Denmark (4):
  - "Aalborg Universitetshospital, Syd Onkologisk Afdeling", Aalborg
  - Rigshospitalet Dpt of Oncology, Copenhagen
  - "Regionshospitalet Herning, Hospitalsenheden Vest Onkologisk Afdeling", Herning
  - "Odense Universitetshospital Department of Oncology", Odense
- France (6):
  - "CHU Jean Minjoz Service d'oncologie médicale", Besançon
  - "CHU Morvan Institut de Cancérologie et d'Hématologie", Brest
  - "Centre de lutte contre le cancer Francois Baclesse UCP Digestif", Caen
  - Hôpital Saint-Antoine Service d'Oncologie Médicale, Paris
  - "Hôpital Européen Georges Pompidou Oncologie Hépatogastroenterologie-oncologie digestive", Paris
  - CHU de Poitiers Pole Régional de Cancérologie, Poitiers
- Germany (4):
  - Onkologische Schwerpunktpraxis Kurfuerstendamm, Berlin
  - Charite Universitätsmedizin Medizinische Klinik m.S. Haemat., Onko., Tumorimmunologie, Berlin
  - Lübecker Onkologische Schwerpunktpraxis im Hochschulstadttei, Lübeck
  - Klinikum der Universität München Campus Großhadern, Medizinische Klinik und Poliklinik III, München
- Hungary (8):
  - Magyar Honvedseg Egeszsegugyi Kozpont Onkologiai Osztaly, Budapest
  - Szent Imre Egyetemi Oktatokorhaz Klinikai Onkologiai Osztaly, Budapest
  - Debreceni Egyetem Orvos es Egeszsegtudomanyi Centrum Onkologiai Intezet, Debrecen
  - Petz Aladar Megyei Oktato Korhaz Onkoradiologiai Osztaly, Győr
  - Bacs-Kiskun Megyei Korhaz Onkoradiologiai Kozpont, Kecskemét
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kp. Onkoterápiás Klinika, Szeged
  - JNSZ Megyei Hetenyi Geza Korhaz es Rendelointezet Megyei Onkologiai Centrum, Szolnok
  - Markusovszky Egyetemi Oktatokorhaz Onkoradiologiai Osztaly, Szombathely
- Italy (9):
  - Azienda Policlinico Universitaria - Presidio Monserrato Oncologia Medica Strada Statale 554 Sestu-Monserrato, Cagliari, Italiy
  - A.O.U. Seconda Universita degli Studi di Napoli U.O.C di Oncologia Medica e di Ematologia Dipartimento Medico di Internistica clinca e sperimentale " F Magrassi - A. Lanzara" Via Sergio Pansisni ,, Napoli
  - Istituto Nazionale Tumori, I.R.C.C.S "Fondazione G Pascale" Struttura Complessa di Oncologia Medica Addominale, Napoli
  - Istituto Oncologico Veneto IOV - IRCCS Unita Operativa Complessa Oncologia Medica 1 Via Gattamelata 64, Padua
  - A.O.U. Pisana-Ospedale Santa Chiara U.O. di Oncologia Medica 2, Pisa
  - Ospedale San Carlo U.O. Oncologia Medica Via Potito Petrone, Ctr Macchia Romana, Potenza
  - Arcispedale Santa Maria Nuova Unità di Oncologia, Reggio Emilia
  - Istituto Clinico Humanita IRCCS Dipartimento di Oncologia Medica ed Ematologia Via Manzoni,, Rozzano (MI)
  - IRCSS Casa Sollievo della Sofferenza Dipartimento Onco-Ematologia Vale Cappuccini 1, San Giovanni Rotondo
- Poland (7):
  - Przychodnia Lekarska "KOMED", Konin
  - SP ZOZ Szpital Uniwersytecki w Krakowie Oddzial Kliniczny Onkologii, Krakow
  - Opolskie Centrum Onkologii im. Tadeusza Koszarowskiego Oddzial Onkologii Klinicznej, Opole
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Slupsku Sp. z o.o., Słupsk
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie Państwowy Instytut Badawczy Klinika Onkologii i Radioterapii, Warsaw
  - Wojskowy Instytut Medyczny Klinika Onkologii, Warsaw
  - Centralny Szpital Kliniczny MSWiA Oddział Radioterapii i Onkologii, Warzszawa
- Pan American Center for Oncology Trials, LLC, Río Piedras, Porto RICO, Puerto Rico
- Russia (12):
  - Arkhangelsk Clinical Oncology Dispensary chemotherapy department, Arkhangelsk
  - Clinical Oncology Dispensary No.1 Chemotherapy Department, Krasnodar
  - Russian Cancer Research Center n.a. NN Blokhin Clinical Pharmacology and Chemotherapy, Moscow
  - University Headache Clinic Outpatient oncology clinic, Moscow
  - Moscow City Oncology Hospital # 62 chemotherapy department, Moscow Region
  - Omsk Clinical Oncologic Dispensary Chemotherapy, Omsk
  - Scientific Centre for Specialized Medical Care (oncological) Chemotherapy, Saint Petersburg
  - National Medical Research Center of Oncology N.N. Petrova, Saint Petersburg
  - Saint Petersburg City Oncology Clilnic, Saint Petersburg
  - Multidisciplinary clinic "Reaviz, Samara
  - Oncology dispensary No.2 Oncology department, Sochi
  - SBIH of YR "Clinical oncology hospital chemotherapy department", Yaroslavl
- Spain (10):
  - "H. Valle de Hebrón Servicio de Oncología - (VHIR)", Barcelona
  - "Hospital de la Santa Creu I Sant Pau Oncología Medica", Barcelona
  - "Hospital Uni. Reina Sofía - Hospital Provincial Departamento de Oncología Médica", Córdoba
  - "INSTITUTO CATALAN DE ONCOLOGÍA - ICO Oncología Médica", L'Hospitalet de Llobregat
  - "Hospital Universitario Ramón y Cajal Servicio de Oncologia Médica", Madrid
  - "HOSPITAL 12 DE OCTUBRE Servicio Oncología Médica", Madrid
  - "Hospital Universitario Marqués de Valdecilla oncología medica", Santander
  - H.VIRGEN DEL ROCIO Servicio de Oncología Médica, Seville
  - H. GENERAL DE VALENCIA Servicio de Oncología Médica, Valencia
  - Hospital Universitario Miguel Servet Edif. de maternidad planta 8. Servicio de Oncología Médical, Zaragoza
- Ukraine (8):
  - Kyiv City Clinical Oncological Centre, Kiev, Ukrain
  - Cherkasy Regional Oncological Dispensary Regional Clinical Oncological Centre, Cherkassy
  - "MI ""Dnipropetrovsk City Multi-field Clinical Hospital #4"" Department of Oncology", Dnipro
  - LLC Ukrainian Center of Tomotherapy "Tomoclinic", Chemoteraphy Department, Kropyvnytskyi
  - National Institute of Cancer Abdominal Oncology Department, Kyiv
  - Medical Center n.a. Acad. Spizhenko "Syber Clinic Spizhenko"" Department of Oncology, Kyiv
  - "Clinical and diagnostic Centre of Medics-rey Inter. Group LLC Hospital of Israeli Oncology "LISOD", Kyiv
  - Podillia Regional Oncology Centre Chemotherapy Department, Vinnitsya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Prager GW, Taieb J, Fakih M, Ciardiello F, Van Cutsem E, Elez E, Cruz FM, Wyrwicz L, Stroyakovskiy D, Papai Z, Poureau PG, Liposits G, Cremolini C, Bondarenko I, Modest DP, Benhadji KA, Amellal N, Leger C, Vidot L, Tabernero J; SUNLIGHT Investigators. Trifluridine-Tipiracil and Bevacizumab in Refractory Metastatic Colorectal Cancer. N Engl J Med. 2023 May 4;388(18):1657-1667. doi: 10.1056/NEJMoa2214963. PMID 37133585
- [Derived] Prager GW, Taieb J, Fakih M, Ciardiello F, Van Cutsem E, Elez E, Wyrwicz L, Stroyakovskiy D, Liposits G, Bondarenko I, Modest DP, Amellal N, Tabernero J; SUNLIGHT Investigators. Plain language summary of SUNLIGHT: trifluridine/tipiracil and bevacizumab for refractory metastatic colorectal cancer. Future Oncol. 2024;20(36):2823-2832. doi: 10.1080/14796694.2024.2366100. Epub 2024 Jul 2. PMID 38953855

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 99 active sites in 13 countries. A total of 659 participants were screened, of which 492 participants were randomized and treated.
Pre-assignment Details: Randomization (1:1 ratio): stratified by geographic region (North America, European Union, Rest of the World), time since 1st metastasis diagnosis (less than [<] 18 months, greater than or equal to [>=] 18 months) and rat sarcoma virus status (wild-type, mutant). Primary analysis of overall survival as primary outcome measure was completed with cutoff date of July 19, 2022; no efficacy analysis was conducted after this cutoff and participants were continued to be followed for safety analysis.
Groups:
- Trifluridine/Tipiracil + Bevacizumab: Participants were administered 35 milligrams per square meter per dose (mg/m²/dose) trifluridine/tipiracil (FTD/TPI) orally twice a day (BID), within 1 hour after completion of morning and evening meals, 5 days on (Day 1 to 5 and Day 8 to 12) with 2 days off (Day 6 to 7 and Day 13 to 14), over 2 weeks, followed by a 14-day rest; with bevacizumab (5 milligrams per kilogram [mg/kg], intravenous [IV] infusion administered every 2 weeks (Day 1 and Day 15). This treatment cycle was repeated every 4 weeks.
Period: Overall Study
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil
Started | 246 | 246
Completed | 0 | 0
Not Completed | 246 | 246
Not completed — Switched to marketed drug | 32 | 4
Not completed — Radiological Progressive Disease | 145 | 146
Not completed — Clinical Progressive Disease | 20 | 20
Not completed — Radiological And Clinical Progressive Disease | 26 | 52
Not completed — Adverse Event | 16 | 16
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 5 | 8

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants to whom a therapeutic unit was randomly assigned using Interactive Web Response System (IWRS). Participants were analyzed in the arm they were assigned by randomization.
Groups:
- Trifluridine/Tipiracil + Bevacizumab: Participants were administered 35 mg/m²/dose FTD/TPI orally BID, within 1 hour after completion of morning and evening meals, 5 days on (Day 1 to 5 and Day 8 to 12) with 2 days off (Day 6 to 7 and Day 13 to 14), over 2 weeks, followed by a 14-day rest; with bevacizumab 5 mg/kg, IV infusion administered every 2 weeks (Day 1 and Day 15). This treatment cycle was repeated every 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil | Total
Number analyzed (Participants) | 246 | 246 | 492
Age, Continuous [Median (Full Range); unit: years] | 62.00 [20.0 to 84.0] | 64.00 [24.0 to 90.0] | 63.00 [20.0 to 90.0]
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 146 | 129 | 275
  From 65-84 years | 100 | 116 | 216
  85 years and over | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 112 | 236
  Male | 122 | 134 | 256
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 215 | 220 | 435
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 26 | 22 | 48

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival defined as the observed time elapsed between the date of randomization and the date of death due to any cause. The primary estimand of interest was defined to assess the effect of the randomized treatments on the survival duration in all participants regardless of whether or not intercurrent events had occurred (treatment policy strategy). Analysis was performed using Kaplan- Meier method.
Time Frame: From date of randomization to the death due to any cause or cut-off date, whichever comes first (maximum duration: up to 20 months)
Population: Analysis was performed on FAS population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil
Number analyzed (Participants) | 246 | 246
months | 10.78 [9.36 to 11.83] | 7.46 [6.34 to 8.57]
Statistical Analysis 1: Comparison: Trifluridine/Tipiracil + Bevacizumab vs Trifluridine/Tipiracil; Overall Survival Median analysis: The primary estimand was defined to assess the effect of the randomized treatments on the survival duration in all participants regardless of whether or not intercurrent events had occurred (treatment policy strategy); Test type: Superiority; p < 0.001, Stratified log-rank test — Stratified log-rank test, with a target p-value < 0.025 for level of significance; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.49 to 0.77] — Hazard ratio and 95% confidence interval was estimated with stratified Cox proportional hazard model

2. Primary Outcome: Survival Probability at 6 Months
Description: Overall survival defined as the observed time elapsed between the date of randomization and the date of death due to any cause. The primary estimand of interest was defined to assess the effect of the randomized treatments on the survival duration in all participants regardless of whether or not intercurrent events had occurred (treatment policy strategy). Analysis was performed using Kaplan- Meier method. In this outcome measure, data of survival probability at 6 months was reported.
Time Frame: From date of randomization until 6 months post treatment
Population: Analysis was performed on FAS population.
Measure: Number (95% Confidence Interval); unit: probability of participants
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil
Number analyzed (Participants) | 246 | 246
probability of participants | 0.77 [0.72 to 0.82] | 0.61 [0.55 to 0.67]

3. Primary Outcome: Survival Probability at 12 Months
Description: Overall survival defined as the observed time elapsed between the date of randomization and the date of death due to any cause. The primary estimand of interest was defined to assess the effect of the randomized treatments on the survival duration in all participants regardless of whether or not intercurrent events had occurred (treatment policy strategy). Analysis was performed using Kaplan- Meier method. In this outcome measure, data of survival probability at 12 months was reported.
Time Frame: From date of randomization until 12 months post treatment
Population: Analysis was performed on FAS population.
Measure: Number (95% Confidence Interval); unit: probability of participants
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil
Number analyzed (Participants) | 246 | 246
probability of participants | 0.43 [0.36 to 0.49] | 0.30 [0.24 to 0.36]

4. Primary Outcome: Survival Probability at 18 Months
Description: Overall survival defined as the observed time elapsed between the date of randomization and the date of death due to any cause. The primary estimand of interest was defined to assess the effect of the randomized treatments on the survival duration in all participants regardless of whether or not intercurrent events had occurred (treatment policy strategy). Analysis was performed using Kaplan- Meier method. In this outcome measure, data of survival probability at 18 months was reported.
Time Frame: From date of randomization until 18 months post treatment
Population: Analysis was performed on FAS population.
Measure: Number (95% Confidence Interval); unit: probability of participants
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil
Number analyzed (Participants) | 246 | 246
probability of participants | 0.28 [0.19 to 0.37] | 0.15 [0.09 to 0.22]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time elapsed between the date of randomisation and the date of radiological tumour progression as per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) assessed by investigator, or death (from any cause), whichever comes first. Progressive Disease (PD) as per RECIST 1.1: at least a 20 percent (%) increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions. Analysis was performed by Kaplan-Meier method.
Time Frame: From randomization to the date of radiological tumour progression or death due to any cause or data cut-off date whichever comes first (i.e., up to 20 months)
Population: Analysis was performed on FAS population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil
Number analyzed (Participants) | 246 | 246
months | 5.55 [4.50 to 5.88] | 2.40 [2.07 to 3.22]
Statistical Analysis 1: Comparison: Trifluridine/Tipiracil + Bevacizumab vs Trifluridine/Tipiracil; PFS Median analysis: A hierarchical testing method was used to control type I error and handle key secondary endpoint analysis. When the primary outcome measure significant testing was then performed sequentially on the key secondary outcome measure. statistically significant at 0.05 level; Test type: Superiority; p < 0.001, Stratified log-rank test — Stratified log-rank test, with a target p-value < 0.025 for level of significance; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.36 to 0.54] — Hazard ratio and 95% confidence interval was estimated with stratified Cox proportional hazard model

6. Secondary Outcome: Probability of Participants With Progression Free Survival at 3, 6, 9 and 12 Months
Description: PFS was defined as the time elapsed between the date of randomisation and the date of radiological tumour progression as per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) assessed by investigator, or death (from any cause), whichever comes first. Progressive Disease (PD) as per RECIST 1.1: at least a 20 percent (%) increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions. Analysis was performed by Kaplan-Meier method. In this outcome measure, data of PFS at 3 months was reported.
Time Frame: From randomization until 3, 6, 9, and 12 months post treatment
Population: Analysis was performed on FAS population.
Measure: Number (95% Confidence Interval); unit: probability of participants
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil
Number analyzed (Participants) | 246 | 246
probability of participants
  At 3 Months | 0.73 [0.67 to 0.78] | 0.45 [0.39 to 0.51]
  At 6 Months | 0.43 [0.37 to 0.49] | 0.16 [0.11 to 0.21]
  At 9 Months | 0.28 [0.22 to 0.34] | 0.05 [0.03 to 0.09]
  At 12 Months | 0.16 [0.12 to 0.21] | 0.01 [0.00 to 0.03]

7. Secondary Outcome: Overall Response Rate (ORR)
Description: Objective response was defined as percentage of participants who achieved complete response (CR) or partial response (PR) according to the RECIST version 1.1 and using investigator's tumour assessment. As per RECIST 1.1, CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum diameters.
Time Frame: From the date of randomization to the date of documentation of progression or death due to any cause or data cut-off, whichever occurred first (i.e., up to 20 months)
Population: Analysis was performed on FAS population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil
Number analyzed (Participants) | 246 | 246
percentage of participants | 6.10 [3.45 to 9.86] | 1.22 [0.25 to 3.52]

8. Secondary Outcome: Percentage of Participants With Disease Control
Description: Disease control is defined as percentage of participants who achieved CR or PR, or stable disease (SD) as per RECIST 1.1 and using investigator's tumour assessment from the date of randomization to until disease progression or death due to any cause. As per RECIST 1.1, CR: disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least a 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters. PD: at least 20% increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions.
Time Frame: From randomization to the date of first documented tumor progression, death due to any cause or data cut-off date whichever comes first (i.e., up to 20 months)
Population: Analysis was performed on FAS population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil
Number analyzed (Participants) | 246 | 246
percentage of participants | 69.51 [63.35 to 75.2] | 41.87 [35.63 to 48.31]

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. Serious adverse events (SAEs) was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as AEs that developed, worsened or became serious during the TEAE period (time from the first dose of study treatment up to 30 days after the last dose of study treatment). TEAEs included both SAEs and non-SAEs.
Time Frame: From baseline (Cycle 1 Day 1) up to 30 days after the last dose of study drug (i.e., up to 30.7 months)
Population: Analysis was performed on safety set which included all participants who had taken at least one dose of investigational medicinal products and were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil
Number analyzed (Participants) | 246 | 246
Participants
  TEAE | 241 | 241
  TESAE | 66 | 79

10. Secondary Outcome: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30): Time to Definitive Deterioration of >=10 Points in Sub-scale Scores - Kaplan-Meier Analysis
Description: EORTC QLQ-C30: 30 item questionnaires with 5 multi-item functional subscales (physical, role, cognitive, emotional, social functioning), 3 multi-item symptom scales (fatigue, nausea/vomiting, and pain), global health/quality of life (QOL) subscale and 6 single items assessing other cancer related symptoms (dyspnea, sleep disturbance, appetite, diarrhea, constipation and financial impact of cancer). It employed twenty-eight 4-point Likert scales with responses from "not at all" to "very much" and GHS/QoL, scored on scale of 1 (very poor) to 7 (excellent). All scales are transformed from raw scores to linear scales ranging 0 to 100. Higher score for functional & GHS/QoL = higher level of functioning, & higher score for symptoms scales = higher symptom burden. Time to definitive >=10 points deterioration: time from date of randomization to first deterioration in QoL score >=10 points compared to baseline with no later improvement or death due to any cause. Kaplan-Meier method was used.
Time Frame: Date of randomization to first deterioration in QoL score >=10 points or death due to any cause, which ever occurred first (i.e., up to 20 months)
Population: Analysis was performed on FAS population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil
Number analyzed (Participants) | 121 | 155
months
  Physical functioning: number analyzed (Participants) | 108 | 149
  Physical functioning | 8.97 [8.15 to 11.83] | 4.50 [3.71 to 5.62]
  Role functioning: number analyzed (Participants) | 113 | 147
  Role functioning | 8.57 [7.49 to 10.94] | 4.40 [3.78 to 5.06]
  Emotional functioning: number analyzed (Participants) | 97 | 128
  Emotional functioning | 9.95 [8.51 to 12.12] | 5.85 [4.70 to 6.60]
  Cognitive functioning: number analyzed (Participants) | 101 | 132
  Cognitive functioning | 9.36 [8.34 to 12.25] | 4.73 [4.07 to 6.11]
  Social functioning: number analyzed (Participants) | 109 | 137
  Social functioning | 8.97 [7.85 to 11.86] | 4.93 [4.14 to 5.88]
  Fatigue: number analyzed (Participants) | 121 | 149
  Fatigue | 8.21 [6.11 to 9.95] | 4.04 [3.19 to 4.83]
  Nausea and vomiting: number analyzed (Participants) | 104 | 136
  Nausea and vomiting | 9.36 [8.51 to 11.86] | 5.06 [4.27 to 6.31]
  Pain: number analyzed (Participants) | 117 | 155
  Pain | 8.57 [6.96 to 10.41] | 4.34 [3.29 to 5.16]
  Dyspnoea: number analyzed (Participants) | 94 | 131
  Dyspnoea | 9.36 [8.54 to 12.25] | 5.65 [4.40 to 6.60]
  Insomnia: number analyzed (Participants) | 96 | 129
  Insomnia | 9.36 [8.54 to 12.25] | 5.75 [4.70 to 6.80]
  Appetite loss: number analyzed (Participants) | 120 | 144
  Appetite loss | 8.34 [6.70 to 10.94] | 4.66 [3.94 to 6.04]
  Constipation: number analyzed (Participants) | 100 | 128
  Constipation | 9.46 [8.34 to 12.12] | 5.55 [4.63 to 6.67]
  Diarrhoea: number analyzed (Participants) | 94 | 125
  Diarrhoea | 10.41 [8.84 to 14.49] | 5.52 [4.70 to 6.60]
  Financial difficulties: number analyzed (Participants) | 100 | 126
  Financial difficulties | 9.36 [8.34 to 12.12] | 6.11 [5.06 to 6.93]

11. Secondary Outcome: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30): Time to Definitive Deterioration of >=10 Points in the Global Health Status Score - Kaplan-Meier Analysis
Description: EORTC QLQ-C30: 30 item questionnaires composed of 5 multi-item functional subscales (physical, role, cognitive, emotional, social functioning), 3 multi-item symptom scales (fatigue, nausea/vomiting, and pain), global health/QOL subscale and 6 single items assessing other cancer related symptoms (dyspnea, sleep disturbance, appetite, diarrhea, constipation and financial impact of cancer). It employed twenty-eight 4-point Likert scales with responses from "not at all" to "very much" and GHS/QoL, scored on scale of 1 (very poor) to 7 (excellent). All scales are transformed from raw scores to linear scales ranging 0 to 100. Higher score for functional & GHS/QoL = higher level of functioning, & higher score for symptoms scales = higher symptom burden. Time to definitive >=10 points deterioration: time from date of randomization to the first deterioration in QoL score >=10 points compared to baseline with no later improvement or death due to any cause. Kaplan-Meier method was used.
Time Frame: as for outcome 10
Population: Analysis was performed on FAS population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil
Number analyzed (Participants) | 120 | 141
months | 8.54 [7.49 to 10.94] | 4.70 [4.01 to 5.78]

12. Secondary Outcome: Change From Baseline in European Quality of Life Group Questionnaire With 5 Dimensions and 5 Levels Per Dimension (EQ-5D-5L): Health State Utility Index Value at Specified Timepoints
Description: The EQ-5D-5L is a standardized measure of health status that provides a general assessment of health utility and consist in 2 sections a descriptive system comprising 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and Visual Analog Scale (VAS). Each dimension has a 5-level response: no problems, slight problems, moderate problems, severe problems, and extreme problems. Response options are measured with a 5-point Likert scale. The 5D-5L systems are converted into a single index utility score between 0 to 1, where higher score indicates a better health state and lower score indicate worse health state.
Time Frame: Baseline, Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6, Cycle 7, Cycle 8, Cycle 9, Cycle 10, Cycle 11, Cycle 12, Cycle 13 and Cycle 14
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil
Number analyzed (Participants) | 201 | 207
score on a scale
  Cycle 1 | 0.004 (0.125) | 0.001 (0.163)
  Cycle 2: number analyzed (Participants) | 196 | 182
  Cycle 2 | -0.003 (0.114) | -0.030 (0.153)
  Cycle 3: number analyzed (Participants) | 165 | 101
  Cycle 3 | -0.014 (0.107) | 0.002 (0.188)
  Cycle 4: number analyzed (Participants) | 146 | 81
  Cycle 4 | -0.016 (0.111) | -0.014 (0.209)
  Cycle 5: number analyzed (Participants) | 114 | 48
  Cycle 5 | -0.003 (0.101) | 0.004 (0.120)
  Cycle 6: number analyzed (Participants) | 98 | 39
  Cycle 6 | -0.010 (0.112) | -0.003 (0.094)
  Cycle 7: number analyzed (Participants) | 74 | 24
  Cycle 7 | -0.007 (0.078) | 0.002 (0.105)
  Cycle 8: number analyzed (Participants) | 68 | 17
  Cycle 8 | -0.016 (0.097) | -0.028 (0.109)
  Cycle 9: number analyzed (Participants) | 51 | 10
  Cycle 9 | -0.024 (0.149) | 0.032 (0.085)
  Cycle 10: number analyzed (Participants) | 43 | 8
  Cycle 10 | -0.003 (0.094) | 0.018 (0.106)
  Cycle 11: number analyzed (Participants) | 33 | 6
  Cycle 11 | -0.008 (0.105) | 0.008 (0.104)
  Cycle 12: number analyzed (Participants) | 26 | 4
  Cycle 12 | -0.025 (0.113) | 0.030 (0.039)
  Cycle 13: number analyzed (Participants) | 18 | 1
  Cycle 13 | -0.037 (0.112) | 0.015
  Cycle 14: number analyzed (Participants) | 11 | 1
  Cycle 14 | -0.034 (0.062) | 0.016

13. Secondary Outcome: Change From Baseline in European Quality of Life Working Group Health Status Measure 5 Dimensions, 5 Levels (EQ-5D-5L) Score: Visual Analogic Scale (VAS) at Specified Timepoints
Description: The EQ-5D-5L is a standardized measure of health status that provides a general assessment of health utility and consist of 2 sections; descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and a VAS. The VAS records the respondent's self-rated health on a 20 centimeter (cm) vertical VAS; the scale went from 0 (worst imaginable health state) to 100 (best imaginable health state). This information can be used as a quantitative measure of health as judged by the individual respondents.
Time Frame: as for outcome 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil
Number analyzed (Participants) | 201 | 207
score on a scale
  Cycle 1 | 2.095 (16.256) | 0.058 (15.749)
  Cycle 2: number analyzed (Participants) | 196 | 182
  Cycle 2 | 0.852 (15.696) | -4.242 (18.302)
  Cycle 3: number analyzed (Participants) | 165 | 101
  Cycle 3 | 0.297 (17.618) | -1.604 (15.729)
  Cycle 4: number analyzed (Participants) | 146 | 81
  Cycle 4 | -0.521 (18.177) | -3.247 (17.769)
  Cycle 5: number analyzed (Participants) | 114 | 48
  Cycle 5 | 1.904 (16.908) | -1.271 (16.738)
  Cycle 6: number analyzed (Participants) | 98 | 39
  Cycle 6 | 2.786 (16.162) | -3.513 (18.602)
  Cycle 7: number analyzed (Participants) | 74 | 24
  Cycle 7 | 1.500 (16.730) | -2.708 (16.573)
  Cycle 8: number analyzed (Participants) | 68 | 17
  Cycle 8 | 0.221 (15.635) | -0.353 (16.328)
  Cycle 9: number analyzed (Participants) | 51 | 10
  Cycle 9 | -1.745 (14.085) | 3.400 (11.928)
  Cycle 10: number analyzed (Participants) | 43 | 8
  Cycle 10 | -1.953 (13.991) | -4.500 (25.785)
  Cycle 11: number analyzed (Participants) | 33 | 6
  Cycle 11 | -1.212 (16.328) | 2.833 (16.388)
  Cycle 12: number analyzed (Participants) | 26 | 4
  Cycle 12 | 2.385 (13.674) | 8.000 (15.188)
  Cycle 13: number analyzed (Participants) | 18 | 1
  Cycle 13 | -2.056 (15.757) | 13.000
  Cycle 14: number analyzed (Participants) | 11 | 1
  Cycle 14 | 0.545 (15.952) | 13.000

ADVERSE EVENTS:
Time Frame: Serious AEs and Other AEs: From baseline (Cycle 1 Day 1) up to 30 days after the last dose of study drug (i.e., up to 30.7 months); All-cause mortality: from baseline (Cycle 1 Day 1) up to end of the study (i.e., up to 33.6 months)
Description: Analysis was performed on safety set population which included all participants who took at least one dose of FTD/TPI and were analyzed according to the treatment actually received. Reported serious AEs and other AEs were treatment-emergent AEs that developed, worsened or became serious from baseline (Cycle 1 Day 1) up to 30 days after the last dose of the study drug.
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Trifluridine/Tipiracil
All-Cause Mortality (participants affected / at risk) | 208/246 | 224/246
Serious Adverse Events (participants affected / at risk) | 66/246 | 79/246
Other Adverse Events (participants affected / at risk) | 241/246 | 241/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trifluridine/Tipiracil + Bevacizumab (N=246) | Trifluridine/Tipiracil (N=246)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 11
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0
Asthenia (General disorders) | 2 | 0
Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 3
Multiple organ dysfunction syndrome (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Death (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Psychomotor retardation (Psychiatric disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Gastrointestinal stoma output decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Diplegia (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 6
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 9 | 5
Vomiting (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Ascites (Gastrointestinal disorders) | 1 | 2
Ileus (Gastrointestinal disorders) | 1 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 2
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 3 | 0
Jaundice (Hepatobiliary disorders) | 1 | 5
Cholangitis (Hepatobiliary disorders) | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 2 | 0
Biliary dilatation (Hepatobiliary disorders) | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 5
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 2
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Prerenal failure (Renal and urinary disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
COVID-19 (Infections and infestations) | 5 | 6
Septic shock (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 2
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 1
Abdominal sepsis (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Intestinal sepsis (Infections and infestations) | 1 | 0
Paracancerous pneumonia (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 0 | 2
Abdominal infection (Infections and infestations) | 0 | 1
Bacterial prostatitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Small intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Neutrophil count increased (Investigations) | 0 | 1
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trifluridine/Tipiracil + Bevacizumab (N=246) | Trifluridine/Tipiracil (N=246)
Neutrophil count decreased (Investigations) | 34 | 18
Platelet count decreased (Investigations) | 24 | 6
Alanine aminotransferase increased (Investigations) | 20 | 14
Aspartate aminotransferase increased (Investigations) | 20 | 14
Weight decreased (Investigations) | 23 | 12
Blood bilirubin increased (Investigations) | 16 | 14
Hypertension (Vascular disorders) | 26 | 5
Headache (Nervous system disorders) | 21 | 9
Neutropenia (Blood and lymphatic system disorders) | 153 | 126
Anaemia (Blood and lymphatic system disorders) | 79 | 80
Thrombocytopenia (Blood and lymphatic system disorders) | 44 | 29
Leukopenia (Blood and lymphatic system disorders) | 19 | 21
Asthenia (General disorders) | 61 | 58
Fatigue (General disorders) | 54 | 41
Pyrexia (General disorders) | 15 | 14
Nausea (Gastrointestinal disorders) | 95 | 69
Diarrhoea (Gastrointestinal disorders) | 54 | 47
Vomiting (Gastrointestinal disorders) | 51 | 36
Abdominal pain (Gastrointestinal disorders) | 31 | 27
Constipation (Gastrointestinal disorders) | 28 | 28
Stomatitis (Gastrointestinal disorders) | 29 | 10
Abdominal pain upper (Gastrointestinal disorders) | 23 | 11
Proteinuria (Renal and urinary disorders) | 15 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 13
Decreased appetite (Metabolism and nutrition disorders) | 55 | 39
COVID-19 (Infections and infestations) | 24 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-12-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT04737187/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT04737187/SAP_001.pdf